CLINICAL TRIAL: NCT03879460
Title: The Evaluation of Safety and Tolerance of Commercially Available Naltrexone Administered Daily - Assessment for CBRN Operations
Acronym: TEST CANADA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Timothy Smith (Other Government)
Responsible Party: Sponsor-Investigator, Timothy Smith, Regulatory & Product Development Specialist, Canadian Department of National Defence
Organization: Canadian Department of National Defence (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-044
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Opioid Intoxication
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Open label safety assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental): Open label
  Interventions: Drug: Naltrexone Hydrochloride

INTERVENTIONS:
Drug: Naltrexone Hydrochloride — 50 mg per os naltrexone hydrochloride

SUMMARY:
The objective of this study is to evaluate the tolerance and safety of naltrexone while performing military specific tasks, and to assess plasma concentrations following naltrexone, administered orally at 50 mg per day for 7 days. The physical and mental/cognitive performance assessments will be conducted at various times prior, during and following drug administration. Daily blood draws will also be taken to assess blood levels of naltrexone and active metabolites for correlation to performance parameters associated with the Military Skill & Tasked Based Fitness Test.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant
* between 18 and 55 years;
* Body weight with a BMI range of 18.5 to 27.0 [or weight within 15% of ideal weight for subject's height and frame (to be based on Metropolitan Life Insurance Company weight tables);
* Healthy, with normal findings in the physical examination and vital signs (BP between 100-140/60-90 mmHg, HR between 60 to 90 beats/min, respiration between 12 to 24 breaths/min, SpO2 >90% breathing room air) and no clinically-significant findings in a 12-lead electrocardiogram;
* No clinical laboratory values outside of the laboratory normal reference range, unless the investigator determines them to be not clinically significant;
* Non-smoking (i.e. having no history of tobacco, or other substance, smoking for greater than or equal to 12 months, and not having smoked within the past year by self-report);
* Negative tests for smoking tobacco (urine cotinine test), alcohol (urine test), hepatitis B- surface antigen, hepatitis C antibody, tuberculin skin-prick test at screening;
* Negative urine screen for drugs of abuse;
* Willing and able to communicate well with the investigator and clinic staff, comply with the study procedure and schedule, and provide written informed consent;
* Able to understand the requirements of the study and sign informed consent;

Exclusion Criteria:

* Current major Axis I psychiatric disorder for which the subject is currently receiving treatment or which would make study compliance an issue;
* Pregnant. A test will be available for prospective participants;
* Breast-feeding women;
* Any condition or therapy which, in the opinion of the investigator, may be significantly worsened by the administration of naltrexone or is likely to interfere with the successful collection of the measures required;
* Acute disease at the time of enrolment (i.e. presence of a moderate or severe illness or infection with or without a fever);
* Febrile illness (oral temperature >37.6º C at the time of drug administration);
* Unstable chronic illnesses;
* Chronic liver, renal or inflammatory bowel disease or collagen vascular disease;
* Clinically significant elevation of ALT and/or AST;
* Active neurological disorder;
* Clinically significant uncontrolled illness or clinically significant surgery within 4 weeks prior to administration of study drug;
* Cancer within the previous 5 years, other than squamous cell or basal cell carcinoma of the skin;
* History of any clinical laboratory abnormality deemed significant by the Principal Investigator;
* History of serious adverse reaction or hypersensitivity to any drug;
* Bleeding tendency resulting from disease or medication rendering blood collection or the injection itself unsafe (use of antiplatelet agents is allowed);
* Coagulation disorders or receiving anticoagulant therapy;
* Inability to tolerate abstinence from caffeine for 24 hours prior to and during the study treatment phase;
* Consumption of alcohol within 24 hours prior to dosing and during the treatment phase;
* History of significant alcohol or drug abuse within one year prior to the screening visit or regular use of alcohol within six months prior to the screening visit (more than 14 units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]);
* Use of soft drugs (such as marijuana) within three months prior to the screening visit or hard drugs (such as cocaine, phencyclidine or crack) within one year prior to the screening visit or positive urine drug screen at screening or positive urine drug screen at screening;
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:

  * 50 mL to 300 mL of whole blood within 30 days;
  * 301 mL to 500 mL of whole blood within 45 days; or
  * more than 500 mL of whole blood within 56 days prior to drug administration.
* Any known or suspected allergy to any constituent of naltrexone;
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal Investigator or Sub-Investigators, contraindicates the subject's participation inthis study;
* Use of any investigational or non-registered drug or participation in an investigational study within 30 days prior to administration of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of naltrexone and its active metabolite, 6 beta naltrexol | Study day 4 - 10

CONTACTS AND LOCATIONS:
Locations (1):
- Department of National Defence, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No